CLINICAL TRIAL: NCT00164502
Title: Limb Loss Self-Management Program: "Promoting Amputee Life Skills"
Brief Title: Limb Loss Self-Management Program
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCBDDD-CCR322981
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2005-09-14 (Estimated); Status verified 2005-09

CONDITIONS: Congenital or Acquired Limb Deficiency

INTERVENTIONS:
Behavioral: Community-based eight session group self-management program

SUMMARY:
The goal of the project is to develop and test the efficacy of a community-based self-management intervention for reducing pain, depression, and improving self-efficacy and function in person with limb loss

DETAILED DESCRIPTION:
Approximately 1.2 million Americans are living with the loss of a limb and the incidence is increasing due to increases in the prevalence of diabetes. Pain, emotional distress, reduced functional abilities are common conditions following limb loss and reduce quality of life. Self-management interventions have been found to be effective in reducing the secondary conditions associated with arthritis and diabetes. Self management uses the principles of cognitive-behavioral therapy including education, self monitoring, problem solving, and skill acquisition.

The goal of the project is to develop and test the efficacy of a community based self management intervention for reducing pain, depression, and improving self efficacy and function in persons with limb loss using a randomized controlled design.

50 groups of 8-10 persons will be randomized to either a control group or a treatment group.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older congenital or acquired limb loss

Exclusion Criteria:

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2003-10; Study Completion 2005-06

PRIMARY OUTCOMES:
self-reported pain
depressed mood
positive affect

SECONDARY OUTCOMES:
increase in activities and participation
improved quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Ellen MacKenzie, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Puget Sound Health Services, Seattle, Washington, United States